CLINICAL TRIAL: NCT05139628
Title: The Impact of Skin Colonization at the Peripheral Venous Catheter Insertion Sites on Catheter Tip Colonization and Catheter Related Blood Stream Infections Among Pediatric Oncology Patients.
Brief Title: Peripheral Venous Catheter Related Blood Stream Infections
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Mohamed Abdel-Hafeez, Assistant Lecturer, Assiut University
Other Study IDs: PVC related BSIs
Record Dates: First submitted 2021-11-18; First posted 2021-12-01 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Catheter-Related Infections
MeSH Terms: conditions — Catheter-Related Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: microbiological identification of samples (skin and blood samples) — Samples will be plated on blood culture plates and will be confirmed biochemically.
  Complete Bacteriological diagnosis will be done. The TTP of each BC bottle will be recorded

SUMMARY:
The aim of this work is to:

1. Study the impact of PIVC skin colonization on catheter tip colonization and the development of CRBSI
2. isolate and identify the organisms causing peripheral venous catheter related blood stream infections in pediatric oncology patients.
3. perform antimicrobial sensitivity testing of isolated organisms.
4. identify the associated risk factors that lead to CRBSIs in such group of patients.

DETAILED DESCRIPTION:
Peripheral intravenous catheters (PIVCs) are small flexible tubes that are vital for the delivery of therapies, such as fluids, drugs, and blood transfusions that are required in up to 70% of hospitalized patients. The PIVC is introduced through the skin into the peripheral veins of the arms, hands, or lower limbs. Despite their relatively short-term use (typically <1 week) they are a potential source of catheter-related bloodstream infections (CRBSIs) implicated in up to 5% of nosocomial bacteremias, with a prevalence of 0.67%-2.4 %. Such infections increase a patient's risk of death, discomfort, and length of hospital stay.

Among pediatric patients with hemato-oncologic disease, intravascular catheter-associated bloodstream infection is the most common cause of bloodstream infections leading to increased mortality and morbidity in such patients. The Mortality rates of bloodstream infections in patients with malignancy are significantly higher than in patients without malignancy. There is a paucity of data on blood stream infections (BSIs) generally amongst paediatric oncology patients in low and middle-income countries, and especially CRBSIs.

Cancer patients are predisposed to BSI for several reasons:

* Alterations in anatomic barriers, both internal and external leading to enhance access of bacteria and fungi to the bloodstream.
* Changes in both cell-mediated and humoral immunity occur related both to the primary tumor and the subsequent treatment.
* Infectious complications in pediatric hematology-oncology patients have been significantly associated with the presence of indwelling catheters.

With most clinical studies focusing on central vascular catheters, infections associated with short peripheral venous catheters have received little attention. While central line-associated bloodstream infections have become an important metric in assessing patient safety, peripheral intravenous catheters (PVCs) remain underappreciated as an intravascular device that is also responsible for catheter-associated bloodstream infections.

Catheter related bloodstream infection (CRBSI) is defined as the presence of bacteremia originating from an intravenous catheter. An estimated 60% of these CRBSIs are associated with the patient's skin flora.The skin is a complex environment that provides greater space for diverse commensal and pathogenic microbes. Catheter colonization occurs by progression of microorganisms to the tip of the catheter along either the inner surface (≥7 days of indwelling time) or the outer surface (<7 days of indwelling time) of the catheter. Even despite skin site decontamination with antiseptic prior to PIVC insertion, bacteria may remain in the hair follicles and lower dermis, and immediately after post insertion catheter, the bacteria begin proliferation. If conditions are particularly favorable, for example moisture from diaphoresis, blood ooze, and numerous hair follicles, bacterial growth becomes faster. Skin bacteria can progressively colonize down the insertion site along the PIVC tract. However, the impact of PIVC skin site colonization on tip colonization and the development of CRBSI has never been investigated comprehensively.

ELIGIBILITY:
Inclusion Criteria:

* The following data will be collected for each patient :
* Age
* Sex
* Type of malignancy
* PIVC location
* Antimicrobial use
* Parenteral nutrition
* Dwell-time
* The reason for removal (eg, treatment complete, PIVC complications, or suspected infection, or routinely (72-96 hours).

Exclusion criteria:

* Patient with existing bloodstream infections.
* or those with any type of infections

Ages: 40 Days to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: • This study will be conducted on pediatric patients admitted to South Egypt Cancer Institute -Assiut University with more than 48hrs of catheter insertion.Patients ( age > 40 days up to 18 years) from both sexes.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Study the impact of Peripheral intravenous catheter skin colonization on catheter tip colonization and the development of Catheter related blood stream infections in pediatric oncology patients and Identify the associated risk factors. | 1 year (Anticipated)
  Isolate and identify the organisms causing CRBSIs and perform antimicrobial sensitivity testing of the isolated organisms.

CONTACTS AND LOCATIONS:
Overall Officials: Nahla M Elsherbiny, Prof. Dr., Study Director — Professor of Medical Microbiology and Immunology Faculty of Medicine - Assiut University; Mona H Abdel-Rahim, A. prof., Study Director — Assistant professor of Medical Microbiology and Immunology

REFERENCES:
- [Background] El-Mahallawy H, Sidhom I, El-Din NH, Zamzam M, El-Lamie MM. Clinical and microbiologic determinants of serious bloodstream infections in Egyptian pediatric cancer patients: a one-year study. Int J Infect Dis. 2005 Jan;9(1):43-51. doi: 10.1016/j.ijid.2003.11.010. PMID 15603994
- [Background] Gaur A, Giannini MA, Flynn PM, Boudreaux JW, Mestemacher MA, Shenep JL, Hayden RT. Optimizing blood culture practices in pediatric immunocompromised patients: evaluation of media types and blood culture volume. Pediatr Infect Dis J. 2003 Jun;22(6):545-52. doi: 10.1097/01.inf.0000069762.44241.0d. PMID 12799512
- [Background] Grice EA, Segre JA. The skin microbiome. Nat Rev Microbiol. 2011 Apr;9(4):244-53. doi: 10.1038/nrmicro2537. PMID 21407241
- [Background] Hughes WT, Armstrong D, Bodey GP, Brown AE, Edwards JE, Feld R, Pizzo P, Rolston KV, Shenep JL, Young LS. 1997 guidelines for the use of antimicrobial agents in neutropenic patients with unexplained fever. Infectious Diseases Society of America. Clin Infect Dis. 1997 Sep;25(3):551-73. doi: 10.1086/513764. PMID 9314442
- [Background] Kong HH. Skin microbiome: genomics-based insights into the diversity and role of skin microbes. Trends Mol Med. 2011 Jun;17(6):320-8. doi: 10.1016/j.molmed.2011.01.013. Epub 2011 Mar 4. PMID 21376666
- [Background] Maki DG, Weise CE, Sarafin HW. A semiquantitative culture method for identifying intravenous-catheter-related infection. N Engl J Med. 1977 Jun 9;296(23):1305-9. doi: 10.1056/NEJM197706092962301. PMID 323710
- [Background] Norgaard M, Larsson H, Pedersen G, Schonheyder HC, Sorensen HT. Haematological malignancies--a predictor of a poor outcome in patients with bacteraemia. J Infect. 2006 Sep;53(3):190-8. doi: 10.1016/j.jinf.2005.10.024. Epub 2005 Dec 13. PMID 16352338
- [Background] Rickard CM, Marsh N, Webster J, Runnegar N, Larsen E, McGrail MR, Fullerton F, Bettington E, Whitty JA, Choudhury MA, Tuffaha H, Corley A, McMillan DJ, Fraser JF, Marshall AP, Playford EG. Dressings and securements for the prevention of peripheral intravenous catheter failure in adults (SAVE): a pragmatic, randomised controlled, superiority trial. Lancet. 2018 Aug 4;392(10145):419-430. doi: 10.1016/S0140-6736(18)31380-1. Epub 2018 Jul 26. PMID 30057103
- [Background] Safdar N, Maki DG. The pathogenesis of catheter-related bloodstream infection with noncuffed short-term central venous catheters. Intensive Care Med. 2004 Jan;30(1):62-7. doi: 10.1007/s00134-003-2045-z. Epub 2003 Nov 26. PMID 14647886
- [Background] Sato A, Nakamura I, Fujita H, Tsukimori A, Kobayashi T, Fukushima S, Fujii T, Matsumoto T. Peripheral venous catheter-related bloodstream infection is associated with severe complications and potential death: a retrospective observational study. BMC Infect Dis. 2017 Jun 17;17(1):434. doi: 10.1186/s12879-017-2536-0. PMID 28623882
- [Background] Soifer NE, Borzak S, Edlin BR, Weinstein RA. Prevention of peripheral venous catheter complications with an intravenous therapy team: a randomized controlled trial. Arch Intern Med. 1998 Mar 9;158(5):473-7. doi: 10.1001/archinte.158.5.473. PMID 9508225
- [Background] Webster J, Osborne S, Rickard CM, Marsh N. Clinically-indicated replacement versus routine replacement of peripheral venous catheters. Cochrane Database Syst Rev. 2019 Jan 23;1(1):CD007798. doi: 10.1002/14651858.CD007798.pub5. PMID 30671926
- [Background] Wisplinghoff H, Seifert H, Wenzel RP, Edmond MB. Current trends in the epidemiology of nosocomial bloodstream infections in patients with hematological malignancies and solid neoplasms in hospitals in the United States. Clin Infect Dis. 2003 May 1;36(9):1103-10. doi: 10.1086/374339. Epub 2003 Apr 14. PMID 12715303